CLINICAL TRIAL: NCT04080492
Title: A Prospective Study to Assess Multi-Domain Patient-Reported Cardiac Quality of Life in Adults With Hypertrophic Cardiomyopathy, Thoracic Aortopathy, and Radiation-Induced Heart Disease: UPLIFT
Brief Title: A Cardiac Disease Quality of Life Study
Acronym: UPLIFT
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Milind Desai, Principal Investigator, The Cleveland Clinic
Other Study IDs: 19-1007
Record Dates: First submitted 2019-09-04; First posted 2019-09-06 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Hypertrophic Obstructive Cardiomyopathy; Thoracic Aortic Dilatation; Heart Disease Caused by Ionising Radiation; Quality of Life
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Hypertrophic Cardiomyopathy: Patients being seen for the first time at the Cleveland Clinic for Hypertrophic Cardiomyopathy.
  Interventions: Other: QOL Survey
- Thoracic Aortic Dilatation: Patients being seen for the first time at the Cleveland Clinic for Thoracic Aortic Dilatation.
  Interventions: Other: QOL Survey
- Radiation Induced Heart Disease: Patients being seen for the first time at the Cleveland Clinic for Radiation-Induced Heart Disease.
  Interventions: Other: QOL Survey

INTERVENTIONS:
Other: QOL Survey — The Cardiac Quality of Life (QOL) survey measures health status in five domains: global, physical, emotional, social, and spiritual health. It also includes questions that assess self-efficacy and resilience. The global section asks about your overall quality of life and satisfaction with health. The physical section asks about symptoms and difficulty performing day-to-day tasks. The emotional section asks about depression, anxiety, and stress. The social section asks about social support and relationships. The spiritual section asks about the spiritual outlook on the burden of heart disease. Responses on a 5-level scale.

SUMMARY:
A prospective, longitudinal, non-comparator, non-randomized observational cohort study to assess the quality of life in adult patients affected by hypertrophic cardiomyopathy and thoracic aortic dilatations who are not amenable to surgery, as well as those affected radiation-induced cardiac disease caused by radiation therapy.

DETAILED DESCRIPTION:
While physicians and patients may be aware of the physical limitations that result from a diagnosis of hypertrophic cardiomyopathy (HCM), thoracic aortic dilatation (TAD) or radiation-induced heart disease (RIHD), there is little research on the impact on quality of life from the limitations imposed with these diagnosis. This study aims to address these unknowns in patients with HCM or TAD as well as radiation-induced heart disease in first-time patients at the Cleveland Clinic. Knowledge gained from this study will provide us the ability for better management of the chronic impacts of the disease by identifying potential risk factors of low quality of life or changes in quality of life over time.

This is a prospective, longitudinal, non-comparator, non-randomized survey study describing QOL outcomes for patients with HCM, TAD, or RIHD. Patients being seen for the first time at the Cleveland Clinic for cardiac disease with no previous or scheduled surgery for HCM or TAD will electronically complete a Cardiac Quality of Life Survey at 3 time points (baseline, 3 month & 9 month). The Cardiac Quality of Life Survey measures the participant's health status in five domains - global, physical, emotional, social, and spiritual - as well as self-efficacy and resilience.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 at time of consent with a confirmed diagnosis of HCM, TAD, and/or RIHD being seen at CC Main Campus for a comprehensive clinical cardiac evaluation (i.e. physician, surgeon, nurse practitioner, geneticist, testing, imaging, etc) to define treatment plan for either diagnosis as per Cleveland Clinic provider.
* Patient or an individual in their social support network has the equipment (phone, computer, tablet) and internet connection to complete the emailed follow-up questionnaires.

Exclusion Criteria:

* Previously had surgery or plans to have surgery (full/mini sternotomy or endovascular) in the next nine months for HCM or TAD.
* Inability or unwillingness to comply with study requirements in the opinion of the investigator.
* Inability to provide informed consent.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will include first-time patients being seen at the Cleveland Clinic whose information will be collected in-person and remotely.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2019-08-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Global domain of Cardiac Quality of Life Survey assessed 9 months after baseline as compared to baseline. | 9 months after baseline visit
  The global domain of the Cardiac Quality of Life Survey assesses global health. Three questions related to 1) Perceived overall quality of life, 2) & 3) Satisfaction with overall health status and with heart health. The Perceived overall quality of life responses range from very poor =1 to very good =5. 2) & 3) Satisfaction responses range from very dissatisfied=1 to very satisfied=5. Total global domain score ranges from 3 to 15 points. The higher the score the less impact the cardiac disease has on quality of life.
Physical domain of Cardiac Quality of Life Survey assessed 9 months after baseline as compared to baseline | 9 months after baseline visit
  The physical domain of the Cardiac Quality of Life Survey assesses physical function. 13 questions. 1) Perception of overall physical health: responses ranging from 1=very poor to 5=very good. 2-6) Difficulty performing day-to-day physical tasks with responses ranging from 1=very easy to 5=very difficult. 7-13) Severity of heart disease symptoms affecting day-to-day physical activities: responses ranging from 1=never to 5=always. Total physical domain score ranges from 13 to 85. The higher the score the less impact the cardiac disease has on physical health.
Emotional domain of Cardiac Quality of Life Survey assessed 3 months after baseline as compared to baseline. | 9 months after baseline visit
  The emotional domain of the Cardiac Quality of Life Survey assesses emotional health. 23 questions. 1) Perception of overall emotional health: responses ranging from 1=very poor to 5=very good. 2) effect of heart disease-related physical limitations on emotional health: responses ranging from 1=always to 5=never. Eight questions asking about anxiety with responses ranging from 1=always to 5=never. Seven questions assessing depression are incorporated with responses ranging from 1=always to 5=never. 19-23) affects from a traumatic event related to their health: responses ranging from 1=always to 5=never. Total emotional domain score ranges from 23 to 115. The higher the score the less impact the cardiac disease has on emotional health.
Social domain of Cardiac Quality of Life Survey assessed 9 months after baseline as compared to baseline. | 9 months after baseline visit
  The social domain of the Cardiac Quality of life survey assesses social interaction and relationships. 10 questions. 1) Overall social interaction and relationships: responses ranging from 1=very poor to 5=very good. 2) Effect of heart disease-related physical limitations on social interaction: responses ranging from 1=always to 5=never. 3-10) Confidence in social interaction with friends and family: responses ranging from 1=always to 5=never. Total social domain score ranges from 10 to 50. The higher the score, the less impact the cardiac disease has on social health.
Spiritual domain of quality of life assessed 9 months after baseline visit as compared to the baseline survey in the outpatient clinic. | 9 months after baseline visit
  The spiritual domain of the Cardiac Quality of life survey assesses attitudes patients have surrounding their faith and health status. 4 questions. One question asks about if one's faith helps in coping with heart-related problems with responses ranging from 1=strongly disagree to 5=strongly agree. Three questions ask about feelings of anger, injustice, and turmoil related to heart disease with responses ranging from 1=strongly agree to 5=strongly disagree. Total spiritual domain score ranges from 4 to 20. The higher the score, the less impact the cardiac disease has on spiritual health.
Self-efficacy assessed 9 months after baseline visit as compared to the baseline survey in the outpatient clinic. | 9 months after baseline visit
  The self-efficacy domain of the Cardiac Quality of Life survey measures self-efficacy as it relates to symptoms of heart disease. Six questions from the Cardiac Self-Efficacy Questionnaire asks about confidence in controlling symptoms, controlling illness, and maintaining daily functioning with responses ranging from 1=strongly disagree to 5=strongly agree. Total self-efficacy score ranges from 6 to 30. The higher the score, the less impact the cardiac disease has on self-efficacy.
Resilience assessed 9 months after baseline visit as compared to the baseline survey in the outpatient clinic. | 9 months after baseline visit
  The resilience domain of the Cardiac Quality of Life survey measures the ability to recover quickly from difficulties. 9 questions asking about adapting to change, coping with stress, overcoming obstacles, and handling unpleasant feelings with responses ranging from 1=strongly disagree to 5=strongly agree. Total resilience score ranges from 9 to 45. The higher the score, more resilient the participant is in facing problems related to cardiac disease.
Impact of heritability of cardiac disease assessed 9 months after baseline visit as compared to the baseline survey in the outpatient clinic. | 9 months after baseline visit
  Patients with thoracic aortic aneurysm or hypertrophic cardiomyopathy were asked questions about how the heritability of their cardiac disease affected their quality of life. 3 questions asking about how heritable cardiac disease affects the health and happiness of family members with responses ranging from 1=always to 5=never. Total score ranges from 3 to 15. The higher the score, the less impact the heritability of the cardiac disease as on the quality of life of the patient.
Impact of radiation-induced heart disease (RIHD) assessed at baseline visit in the outpatient clinic. | Baseline visit
  RIHD patients are asked about radiation therapy history, awareness of risk of RIHD, and impact on QOL. 7 questions. One question asks about time since last radiation therapy, ranging from 1= less than 5 years ago to 5=more than 30years ago. Another asks about time since RIHD diagnosis, ranging from 1=within the past week to 5=more than five years ago. One question asks about the duration of time between the symptoms of RIHD and diagnosis of RIHD with responses ranging from 1= less than 1 month to 5=more than 1 year. One question asks about the awareness of risk of RIHD before radiation therapy with responses ranging from 1=strongly disagree to 5=strongly agree. These four questions were not totaled. Three questions ask about the overall QOL before and after RIHD diagnosis and after treatment for RIHD. Responses ranged from 1=very poor to 5=very good. Total score for this section ranges from 3 to 15 with a higher score indicating RIHD had less of an impact on the overall QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Milind Desai, M. D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States